CLINICAL TRIAL: NCT02515864
Title: A Crossover Study to Assess the Effects of FYU-981 on the QT/QTc Interval in Healthy Male and Female Volunteers
Brief Title: Clinical Pharmacology of FYU-981 (Effect on QT/QTc Interval)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FYU-981-007
Record Dates: First submitted 2015-07-29; First posted 2015-08-05 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Male and Female Volunteers
MeSH Terms: interventions — dotinurad; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- FYU-981 anticipated therapeutic dose (Experimental): Drug: FYU-981, FYU-981 Placebo, Moxifloxacin Placebo (Oral)
  Interventions: Drug: FYU-981; Drug: Placebo; Drug: Moxifloxacin Placebo
- FYU-981 supratherapeutic dose (Experimental): Drug: FYU-981, Moxifloxacin Placebo (Oral)
  Interventions: Drug: FYU-981; Drug: Moxifloxacin Placebo
- Placebo (Placebo Comparator): Drug: FYU-981 Placebo, Moxifloxacin Placebo (Oral)
  Interventions: Drug: Placebo; Drug: Moxifloxacin Placebo
- Moxifloxacin (Active Comparator): Drug: Moxifloxacin, FYU-981 Placebo (Oral)
  Interventions: Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: FYU-981
  Arms: FYU-981 anticipated therapeutic dose; FYU-981 supratherapeutic dose
Drug: Placebo
  Arms: FYU-981 anticipated therapeutic dose; Moxifloxacin; Placebo
Drug: Moxifloxacin
  Arms: Moxifloxacin
Drug: Moxifloxacin Placebo
  Arms: FYU-981 anticipated therapeutic dose; FYU-981 supratherapeutic dose; Placebo

SUMMARY:
A Placebo-controlled, Four Way Crossover Study to Investigate the Effect on QT/QTc Interval of a Single Dose of FYU-981, Compared with Placebo, Using Moxifloxacin as a Positive Control, in Healthy Male and Female Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Japanese adult subjects
* Body mass index: >=18.5 and <27.5

Exclusion Criteria:

* Subjects with any disease or any history of diseases that might be unsuitable for participation in the clinical study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
QT/QTc Interval | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Kanagawa, Japan